CLINICAL TRIAL: NCT03205163
Title: A Phase 1/2a, Open-Label, Dose-Escalation Study to Determine the Safety, Tolerability, and Pharmacokinetics of a Single Intravenous Injection of rFVIIIFc-VWF-XTEN (BIVV001) in Previously Treated Adults With Severe Hemophilia A
Brief Title: A Safety, Tolerability, and Pharmacokinetics Study of a Single Intravenous Injection of Recombinant Coagulation Factor VIII Fc - Von Willebrand Factor - XTEN Fusion Protein (rFVIIIFc-VWF-XTEN) (BIVV001) in Previously Treated Adults With Severe Hemophilia A (EXTEN-A)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: TDU16220; 242HA101 (Other: Bioverativ, a Sanofi company)
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Results first posted 2019-12-02 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; BIVV001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Dose Cohort: Advate 25 IU/kg Then BIVV001 25 IU/kg (Experimental): Participants received a single intravenous (IV) dose of Advate 25 international units per kilogram (IU/kg) on Day 1 of Advate treatment period (3 days) followed by a single IV dose of BIVV001 25 IU/kg in BIVV001 treatment period (BTP) (28 days). Advate treatment period (ATP) consisted of a washout of at least 72 hours which was started from the time of Advate dosing.
  Interventions: Biological: Advate (Low Dose); Biological: BIVV001 (Low Dose)
- High Dose Cohort: Advate 65 IU/kg Then BIVV001 65 IU/kg (Experimental): Participants received a single IV dose of Advate 65 IU/kg on Day 1 of ATP (4 days) followed by a single IV dose of BIVV001 65 IU/kg in BTP (28 days). ATP consisted of a washout of at least 96 hours which was started from the time of Advate dosing.
  Interventions: Biological: Advate (High Dose); Biological: BIVV001 (High Dose)

INTERVENTIONS:
Biological: Advate (Low Dose) — Participants received a single IV low dose of Advate 25 IU/kg.
  Arms: Low Dose Cohort: Advate 25 IU/kg Then BIVV001 25 IU/kg
Biological: Advate (High Dose) — Participants received a single IV high dose of Advate 65 IU/kg.
  Arms: High Dose Cohort: Advate 65 IU/kg Then BIVV001 65 IU/kg
Biological: BIVV001 (Low Dose) — Participants received single IV low dose of BIVV001 25 IU/kg.
  Arms: Low Dose Cohort: Advate 25 IU/kg Then BIVV001 25 IU/kg
Biological: BIVV001 (High Dose) — Participants received single IV high dose of BIVV001 65 IU/kg.
  Arms: High Dose Cohort: Advate 65 IU/kg Then BIVV001 65 IU/kg

SUMMARY:
The primary purpose was to assess the safety and tolerability of a single intravenous (IV) administration of BIVV001 in adult previously treated patients (PTPs) with severe hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Ability of the participant, or his legally authorized representative (e.g., parent or legal guardian) if applicable in accordance with local regulations, to understand the purpose and risks of the study and provide signed and dated informed consent/assent and authorization to use confidential health information in accordance with national and local participant privacy regulations.
* Severe hemophilia A, defined as less than (<) 1 international units per deciliter (IU/dL) (<1 percent [%]) endogenous FVIII at screening as determined by the one-stage clotting assay from the central laboratory. If the initial screening result was greater than or equal to (>=) 1%, then a repeat endogenous FVIII activity level was performed using the one stage clotting assay from the central laboratory. If the repeated result was < 1 IU/dL (<1%), then the participant met this inclusion requirement.
* Previous treatment for hemophilia A, defined as at least 150 documented prior exposure days to any recombinant and/or plasma-derived FVIII and/or cryoprecipitate products at Day 1. Fresh frozen plasma treatment must not be considered in the count for documented exposure days.
* Platelet count >=100,000 cells/ microliter (mcL) at screening (test performed by the central laboratory and reviewed prior to the Day 1 Advate dose).
* A participant known to be human immunodeficiency virus (HIV) antibody positive, either previously documented or identified from screening assessments, must have the following results prior to Day 1 Advate dose: cluster of differentiation 4 (CD4) lymphocyte count greater than (>) 200 cells/millimeter (mm)^3; viral load of <400 copies/mL.

Exclusion Criteria:

Medical History:

* Any concurrent clinically significant major disease that, in the opinion of the Investigator, made the participant unsuitable for enrollment.
* Serious active bacterial or viral infection (other than chronic hepatitis or HIV) present within 30 days of screening.
* Other known coagulation disorder(s) in addition to hemophilia A.
* History of hypersensitivity or anaphylaxis associated with any FVIII product.
* Known or suspected allergy to mice, hamsters, or any ingredient in Advate.
* History of a positive inhibitor test or clinical signs of decreased response to FVIII administrations. Family history of inhibitors not excluded the participant.

Medications and Procedures:

- Current enrollment or participation within 30 days prior to screening in any other investigational study.

Other:

* Inability to comply with study requirements as assessed by the Investigator.
* Other unspecified reasons that, in the opinion of the Investigator or Sponsor, made the participant unsuitable for enrollment.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (7):
  - University of California Los Angeles Medical Center, Los Angeles, California
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Michigan State University, East Lansing, Michigan
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Hemophilia Center of Western PA, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington
- Japan (3):
  - Nara Medical University Hospital, Kashihara-shi, Nara
  - Tokyo Medical University Hospital, Shinjuku-Ku, Tokyo-To
  - Ogikubo Hospital, Tokyo, Tokyo-To

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Konkle BA, Shapiro AD, Quon DV, Staber JM, Kulkarni R, Ragni MV, Chhabra ES, Poloskey S, Rice K, Katragadda S, Fruebis J, Benson CC. BIVV001 Fusion Protein as Factor VIII Replacement Therapy for Hemophilia A. N Engl J Med. 2020 Sep 10;383(11):1018-1027. doi: 10.1056/NEJMoa2002699. PMID 32905674

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Japan and United States between 28 August 2017 to 12 November 2018.
Pre-assignment Details: A total of 16 participants were enrolled, 7 participants to low dose cohort (LDC) and 9 to high dose cohort (HDC).
Groups:
- Low Dose Cohort (LDC): Advate 25 IU/kg Then BIVV001 25 IU/kg: Participants received a single intravenous (IV) dose of Advate 25 International Units per kilogram (IU/kg) on Day 1 of Advate treatment period (ATP) (3 days) followed by a single IV dose of BIVV001 25 IU/kg in BIVV001 treatment period (BTP) (28 days). ATP consisted of a washout of at least 72 hours which was started from the time of Advate dosing.
- High Dose Cohort (HDC): Advate 65 IU/kg Then BIVV001 65 IU/kg: Participants received a single IV dose of Advate 65 IU/kg on Day 1 of ATP (4 days) followed by a single IV dose of BIVV001 65 IU/kg in BTP (28 days). ATP consisted of a washout of at least 96 hours which was started from the time of Advate dosing.
Period: ATP (LDC: 3 Days; HDC: 4 Days)
Arm/Group | Low Dose Cohort (LDC): Advate 25 IU/kg Then BIVV001 25 IU/kg | High Dose Cohort (HDC): Advate 65 IU/kg Then BIVV001 65 IU/kg
Started | 7 | 9
Safety Population | 7 | 9
Completed | 6 | 9
Not Completed | 1 | 0
Not completed — Sponsor Decision | 1 | 0
Period: BTP (LDC: 28 Days; HDC: 28 Days)
Arm/Group | Low Dose Cohort (LDC): Advate 25 IU/kg Then BIVV001 25 IU/kg | High Dose Cohort (HDC): Advate 65 IU/kg Then BIVV001 65 IU/kg
Started | 6 | 9
Safety Population | 6 | 9
Completed | 6 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included all enrolled participants.
Groups:
- LDC: Advate 25 IU/kg Then BIVV001 25 IU/kg: Participants received a single IV dose of Advate 25 IU/kg on Day 1 of ATP (3 days) followed by a single IV dose of BIVV001 25 IU/kg in BTP (28 days). ATP consisted of a washout of at least 72 hours which was started from the time of Advate dosing.
- HDC: Advate 65 IU/kg Then BIVV001 65 IU/kg: Participants received a single IV dose of Advate 65 IU/kg on Day 1 of ATP (4 days) followed by a single IV dose of BIVV001 65 IU/kg in BTP (28 days). ATP consisted of a washout of at least 96 hours which was started from the time of Advate dosing.
- Total: Total of all reporting groups
Arm/Group | LDC: Advate 25 IU/kg Then BIVV001 25 IU/kg | HDC: Advate 65 IU/kg Then BIVV001 65 IU/kg | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (13.81) | 44.0 (11.65) | 39.2 (13.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) and Treatment Emergent Serious Adverse Event (TESAE) During Advate Treatment Period
Description: AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had a causal relationship with the treatment. TEAE is defined as any AE that begins on or after the single dose of Advate but before the single dose of BIVV001. Serious AE (SAE) was defined as any AE resulting in death, immediate risk of death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, or a congenital/anomaly/birth defect, or any other medically important event.
Time Frame: Up to Day 3 for Advate 25 IU/kg; up to Day 4 for Advate 65 IU/kg
Population: Analysis was performed on safety analysis set which included all participants who received at least 1 dose of Advate.
Measure: Count of Participants; unit: Participants
Groups:
- Advate 25 IU/kg: Participants received a single IV dose of Advate 25 IU/kg on Day 1 of ATP (3 days).
- Advate 65 IU/kg: Participants received a single IV dose of Advate 65 IU/kg on Day 1 of ATP (4 days).
Arm/Group | Advate 25 IU/kg | Advate 65 IU/kg
Number analyzed (Participants) | 7 | 9
Participants
  TEAE | 2 | 1
  TESAE | 1 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) and Treatment Emergent Serious Adverse Event (TESAE) During BIVV001 Treatment Period
Description: AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had a causal relationship with the treatment. TEAE is defined as any AE that begins on or after the study treatment (BIVV001) and within 28 days after BIVV001 administration. SAE was defined as any AE resulting in death, immediate risk of death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, or a congenital/anomaly/birth defect, or any other medically important event.
Time Frame: Up to 28 days after BIVV001 administration
Population: Analysis was performed on safety analysis set which included all participants who received at least 1 dose of BIVV001.
Measure: Count of Participants; unit: Participants
Groups:
- BIVV001 25 IU/kg: Participants received a single IV dose of BIVV001 25 IU/kg on Day 1 in BTP (28 days).
- BIVV001 65 IU/kg: Participants received a single IV dose of BIVV001 65 IU/kg on Day 1 in BTP (28 days).
Arm/Group | BIVV001 25 IU/kg | BIVV001 65 IU/kg
Number analyzed (Participants) | 6 | 9
Participants
  TEAE | 3 | 6
  TESAE | 1 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Tests During Advate Treatment Period
Description: Number of Participants with Clinically Significant Abnormalities in Laboratory tests (including hematology, clinical chemistry, urinalysis, and coagulation and thrombosis markers) was reported.
Time Frame: Up to Day 3 for Advate 25 IU/kg; up to Day 4 for Advate 65 IU/kg
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Advate 25 IU/kg | Advate 65 IU/kg
Number analyzed (Participants) | 7 | 9
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Tests During BIVV001 Treatment Period
Description: Number of participants with clinically significant abnormalities (including hematology, clinical chemistry, urinalysis, and coagulation and thrombosis markers) was reported.
Time Frame: Up to 28 days after BIVV001 administration
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | BIVV001 25 IU/kg | BIVV001 65 IU/kg
Number analyzed (Participants) | 6 | 9
Participants | 0 | 0

5. Primary Outcome: Percentage of Participants With Confirmed Inhibitor Development as Measured by the Nijmegen-Modified Bethesda Assay
Description: Development of an inhibitor was defined as a neutralizing antibody value of greater than or equal to (>=) 0.6 Bethesda units per milliliter (BU/mL) identified and confirmed by a second test on an independent sample, collected within 2 to 4 weeks of the first positive sample, with both tests performed by the central laboratory using Nijmegen-modified Bethesda assay.
Time Frame: Up to 28 days after BIVV001 administration
Population: Analysis was performed on safety analysis set.
Measure: Number; unit: percentage of participants
Groups:
- Low Dose Cohort (LDC): Advate 25 IU/kg Then BIVV001 25 IU/kg: Participants received a single IV dose of Advate 25 IU/kg on Day 1 of ATP (3 days) followed by a single IV dose of BIVV001 25 IU/kg in BTP (28 days). ATP consisted of a washout of at least 72 hours which was started from the time of Advate dosing.
- High Dose Cohort (HDC): Advate 65 IU/kg Then BIVV001 65 IU/kg: Participants received a single IV dose of Advate 65 IU/kg on Day 1 of ATP (4 days) followed by a single IV dose of BIVV001 65 IU/kg in BTP (28 days). Advate treatment period consisted of a washout of at least 96 hours which was started from the time of Advate dosing.
Arm/Group | Low Dose Cohort (LDC): Advate 25 IU/kg Then BIVV001 25 IU/kg | High Dose Cohort (HDC): Advate 65 IU/kg Then BIVV001 65 IU/kg
Number analyzed (Participants) | 7 | 9
percentage of participants | 0 | 0

6. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) for Advate and BIVV001 (Low Dose Comparison)
Description: Cmax of Advate and BIVV001 at low dose was assessed and compared based on One-stage activated partial thromboplastin time (aPTT)-based clotting assay.
Time Frame: For Advate: Pre-dose and Post dose at 0.5, 1, 6, 24, 48, and 72 hours; For BIVV001: Pre-dose and Post dose at 0.17, 0.5, 1, 3, 6, 9, 24, 48, 72, 96, 120, 168, and 240 hours
Population: Analysis was performed on pharmacokinetic analysis set (PKAS) which included participants who had adequate blood sample collections (following Advate or BIVV001 administration), to assess key PK parameters, as determined by the PK scientist.
Measure: Geometric Mean (95% Confidence Interval); unit: International unit/deciliter (IU/dL)
Groups:
- Advate 25 IU/kg: Participants received a single IV dose of Advate 25 IU/kg on Day 1 in ATP (3 days).
Arm/Group | Advate 25 IU/kg | BIVV001 25 IU/kg
Number analyzed (Participants) | 7 | 6
International unit/deciliter (IU/dL) | 51.8 [43.3 to 61.9] | 70.1 [49.7 to 98.9]
Statistical Analysis 1: Comparison: Advate 25 IU/kg vs BIVV001 25 IU/kg; Comparison of Advate and BIVV001 was obtained through analyzing log transformed PK parameters using an analysis of variance (ANOVA) model containing participant and treatment as factors. Geometric mean, 95% confidence interval of geometric mean, and geometric mean ratio (GMR) were the exponentiated mean, 95% confidence interval, and difference of means, respectively; Test type: Other; p = 0.032, ANOVA; GMR = 1.35, 95% CI 2-sided [1.04 to 1.77]

7. Secondary Outcome: PK: Maximum Observed Plasma Concentration (Cmax) for Advate and BIVV001 (High Dose Comparison)
Description: Cmax of Advate and BIVV001 at high dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: For Advate: Pre-dose and Post dose at 0.5, 1, 6, 24, 48, and 72 hours; For BIVV001: Pre-dose and Post dose at 0.17, 0.5, 1, 3, 6, 9, 24, 48, 72, 96, 120, 168, 240, 288, and 336 hours
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Groups:
- Advate 65 IU/kg: Participants received a single IV dose of Advate 65 IU/kg on Day 1 in ATP (4 days).
Arm/Group | Advate 65 IU/kg | BIVV001 65 IU/kg
Number analyzed (Participants) | 9 | 8
IU/dL | 138 [117 to 162] | 161 [142 to 183]
Statistical Analysis 1: Comparison: Advate 65 IU/kg vs BIVV001 65 IU/kg; Comparison of Advate and BIVV001 was obtained through analyzing log transformed PK parameters using an ANOVA model containing participant and treatment as factors. Geometric mean, 95% confidence interval of geometric mean, and GMR were the exponentiated mean, 95% confidence interval, and difference of means, respectively; Test type: Other; p < 0.001, ANOVA; GMR = 1.17, 95% CI 2-sided [1.09 to 1.25]

8. Secondary Outcome: PK: Half-Life (t1/2) for Advate and BIVV001 (Low Dose Comparison)
Description: Half-life is defined as time required for the concentration of the drug to reach half of its original value. t1/2 of Advate and BIVV001 at low dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: as for outcome 6
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Advate 25 IU/kg | BIVV001 25 IU/kg
Number analyzed (Participants) | 7 | 6
hours | 9.12 [6.24 to 13.33] | 37.61 [33.28 to 42.50]
Statistical Analysis 1: Comparison: Advate 25 IU/kg vs BIVV001 25 IU/kg; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.001, ANOVA; GMR = 4.13, 95% CI 2-sided [2.94 to 5.79]

9. Secondary Outcome: PK: Half-Life for Advate and BIVV001 (High Dose Comparison)
Description: Half-life is defined as time required for the concentration of the drug to reach half of its original value. t1/2 of Advate and BIVV001 at high dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: as for outcome 7
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Advate 65 IU/kg | BIVV001 65 IU/kg
Number analyzed (Participants) | 9 | 8
hours | 13.15 [10.89 to 15.87] | 42.54 [39.72 to 45.56]
Statistical Analysis 1: Comparison: Advate 65 IU/kg vs BIVV001 65 IU/kg; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.001, ANOVA; GMR = 3.24, 95% CI 2-sided [2.76 to 3.79]

10. Secondary Outcome: PK: Total Body Clearance (CL) for Advate and BIVV001 (Low Dose Comparison)
Description: Clearance is defined as a quantitative measure of the rate at which a drug substance is removed from the body. CL of Advate and BIVV001 at low dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: as for outcome 6
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: milliliter/hour/kilogram (mL/hr/kg)
Arm/Group | Advate 25 IU/kg | BIVV001 25 IU/kg
Number analyzed (Participants) | 7 | 6
milliliter/hour/kilogram (mL/hr/kg) | 3.91 [3.05 to 5.02] | 0.558 [0.411 to 0.757]
Statistical Analysis 1: Comparison: Advate 25 IU/kg vs BIVV001 25 IU/kg; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.001, ANOVA; GMR = 0.143, 95% CI 2-sided [0.118 to 0.172]

11. Secondary Outcome: PK: Total Body Clearance (CL) for Advate and BIVV001 (High Dose Comparison)
Description: Clearance is defined as a quantitative measure of the rate at which a drug substance is removed from the body. CL of Advate and BIVV001 at high dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: as for outcome 7
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/hr/kg
Arm/Group | Advate 65 IU/kg | BIVV001 65 IU/kg
Number analyzed (Participants) | 9 | 8
mL/hr/kg | 3.31 [2.81 to 3.88] | 0.505 [0.436 to 0.586]
Statistical Analysis 1: Comparison: Advate 65 IU/kg vs BIVV001 65 IU/kg; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.001, ANOVA; GMR = 0.153, 95% CI 2-sided [0.138 to 0.170]

12. Secondary Outcome: PK: Volume of Distribution at Steady State (Vss) for Advate and BIVV001 (Low Dose Comparison)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss of Advate and BIVV001 at low dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: as for outcome 6
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: milliliter/kilogram (mL/kg)
Arm/Group | Advate 25 IU/kg | BIVV001 25 IU/kg
Number analyzed (Participants) | 7 | 6
milliliter/kilogram (mL/kg) | 55.9 [51.2 to 61.0] | 34.8 [27.3 to 44.3]
Statistical Analysis 1: Comparison: Advate 25 IU/kg vs BIVV001 25 IU/kg; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.003, ANOVA; GMR = 0.622, 95% CI 2-sided [0.492 to 0.786]

13. Secondary Outcome: PK: Volume of Distribution at Steady State (Vss) for Advate and BIVV001 (High Dose Comparison)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss of Advate and BIVV001 at high dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: as for outcome 7
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | Advate 65 IU/kg | BIVV001 65 IU/kg
Number analyzed (Participants) | 9 | 8
mL/kg | 58.3 [49.8 to 68.2] | 35.0 [29.7 to 41.1]
Statistical Analysis 1: Comparison: Advate 65 IU/kg vs BIVV001 65 IU/kg; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.001, ANOVA; GMR = 0.599, 95% CI 2-sided [0.525 to 0.684]

14. Secondary Outcome: PK: Area Under the Concentration Time Curve (AUC) From Time 0 to Infinity (AUCinfinity) for Advate and BIVV001 (Low Dose Comparison)
Description: AUCinfinity of Advate and BIVV001 at low dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: as for outcome 6
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: hour*international unit/deciliter
Arm/Group | Advate 25 IU/kg | BIVV001 25 IU/kg
Number analyzed (Participants) | 7 | 6
hour*international unit/deciliter | 638 [495 to 822] | 4470 [3280 to 6080]
Statistical Analysis 1: Comparison: Advate 25 IU/kg vs BIVV001 25 IU/kg; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.001, ANOVA; GMR = 7.00, 95% CI 2-sided [5.78 to 8.48]

15. Secondary Outcome: PK: Area Under the Concentration Time Curve From Time 0 to Infinity (AUCinfinity) for Advate and BIVV001 (High Dose Comparison)
Description: AUCinfinity of Advate and BIVV001 at high dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: as for outcome 7
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: hour*international unit/deciliter
Arm/Group | Advate 65 IU/kg | BIVV001 65 IU/kg
Number analyzed (Participants) | 9 | 8
hour*international unit/deciliter | 1960 [1670 to 2310] | 12800 [11100 to 14900]
Statistical Analysis 1: Comparison: Advate 65 IU/kg vs BIVV001 65 IU/kg; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.001, ANOVA; GMR = 6.54, 95% CI 2-sided [5.89 to 7.27]

16. Secondary Outcome: PK: Mean Residence Time (MRT) for Advate and BIVV001 (Low Dose Comparison)
Description: The average time at which the number of absorbed molecules reside in the body, after single-dose administration. MRT of Advate and BIVV001 at low dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: as for outcome 6
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Advate 25 IU/kg | BIVV001 25 IU/kg
Number analyzed (Participants) | 7 | 6
hours | 12.54 [9.82 to 16.01] | 56.93 [49.19 to 65.89]
Statistical Analysis 1: Comparison: Advate 25 IU/kg vs BIVV001 25 IU/kg; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.001, ANOVA; GMR = 4.54, 95% CI 2-sided [3.64 to 5.66]

17. Secondary Outcome: PK: Mean Residence Time (MRT) for Advate and BIVV001 (High Dose Comparison)
Description: The average time at which the number of absorbed molecules reside in the body, after single-dose administration. MRT of Advate and BIVV001 at high dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: as for outcome 7
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Advate 65 IU/kg | BIVV001 65 IU/kg
Number analyzed (Participants) | 9 | 8
hours | 15.66 [14.06 to 17.45] | 67.66 [62.59 to 73.14]
Statistical Analysis 1: Comparison: Advate 65 IU/kg vs BIVV001 65 IU/kg; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.001, ANOVA; GMR = 4.32, 95% CI 2-sided [3.96 to 4.72]

18. Secondary Outcome: PK: Incremental Recovery (IR) for Advate and BIVV001 (Low Dose Comparison)
Description: Incremental Recovery is defined as the increase in the circulating FVIII activity level for one unit (IU) of the FVIII product per kilogram body weight. IR of Advate and BIVV001 at low dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: as for outcome 6
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | Advate 25 IU/kg | BIVV001 25 IU/kg
Number analyzed (Participants) | 7 | 6
IU/dL per IU/kg | 2.0 [1.60 to 2.50] | 2.72 [1.95 to 3.80]
Statistical Analysis 1: Comparison: Advate 25 IU/kg vs BIVV001 25 IU/kg; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.063, ANOVA; GMR = 1.36, 95% CI 2-sided [0.978 to 1.89]

19. Secondary Outcome: PK: Incremental Recovery (IR) for Advate and BIVV001 (High Dose Comparison)
Description: Incremental Recovery is defined as the increase in the circulating FVIII activity level for one unit (IU) of the FVIII product per kilogram body weight. IR of Advate and BIVV001 at high dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: as for outcome 7
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | Advate 65 IU/kg | BIVV001 65 IU/kg
Number analyzed (Participants) | 9 | 8
IU/dL per IU/kg | 2.11 [1.79 to 2.49] | 2.48 [2.18 to 2.82]
Statistical Analysis 1: Comparison: Advate 65 IU/kg vs BIVV001 65 IU/kg; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.001, ANOVA; GMR = 1.18, 95% CI 2-sided [1.10 to 1.26]

20. Secondary Outcome: PK: Time to 1% Above Baseline for FVIII Activity for Advate and BIVV001 (Low Dose Comparison)
Description: Time to 1% activity is the time required from the start of dosing for the FVIII activity to reach 1 IU/dL (1%) above their baseline levels. Time to 1% above baseline for FVIII Activity of Advate and BIVV001 at low dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: as for outcome 6
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Advate 25 IU/kg | BIVV001 25 IU/kg
Number analyzed (Participants) | 7 | 6
hours | 56.97 [49.25 to 65.89] | 260.53 [222.34 to 305.30]
Statistical Analysis 1: Comparison: Advate 25 IU/kg vs BIVV001 25 IU/kg; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.001, ANOVA; GMR = 4.57, 95% CI 2-sided [4.00 to 5.23]

21. Secondary Outcome: PK: Time to 1% Above Baseline for FVIII Activity for Advate and BIVV001 (High Dose Comparison)
Description: Time to 1% activity is the time required from the start of dosing for the FVIII activity to reach 1 IU/dL (1%) above their baseline levels. Time to 1% above baseline for FVIII Activity of Advate and BIVV001 at high dose was assessed and compared based on One-stage aPTT-based clotting assay.
Time Frame: as for outcome 7
Population: Analysis was performed on PKAS.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Advate 65 IU/kg | BIVV001 65 IU/kg
Number analyzed (Participants) | 9 | 8
hours | 78.48 [70.88 to 86.89] | 350.34 [326.61 to 375.81]
Statistical Analysis 1: Comparison: Advate 65 IU/kg vs BIVV001 65 IU/kg; [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.001, ANOVA; GMR = 4.46, 95% CI 2-sided [4.16 to 4.79]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to end of the study (28 days after BIVV001 administration) regardless of seriousness or relationship to investigational product.
Description: Analysis was performed on safety analysis set.
Groups:
- Advate Dose Level: 25 IU/kg: Participants received a single IV dose of Advate 25 IU/kg on Day 1 of ATP (3 days).
- Advate Dose Level: 65 IU/kg: Participants received a single IV dose of Advate 65 IU/kg on Day 1 of ATP (4 days).
- BIVV001 Dose Level: 25 IU/kg: Participants received a single IV dose of BIVV001 25 IU/kg on Day 1 in BTP (28 days).
- BIVV001 Dose Level: 65 IU/kg: Participants received a single IV dose of BIVV001 65 IU/kg on Day 1 in BTP (28 days).
Arm/Group | Advate Dose Level: 25 IU/kg | Advate Dose Level: 65 IU/kg | BIVV001 Dose Level: 25 IU/kg | BIVV001 Dose Level: 65 IU/kg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9 | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/9 | 1/6 | 0/9
Other Adverse Events (participants affected / at risk) | 1/7 | 1/9 | 3/6 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Advate Dose Level: 25 IU/kg (N=7) | Advate Dose Level: 65 IU/kg (N=9) | BIVV001 Dose Level: 25 IU/kg (N=6) | BIVV001 Dose Level: 65 IU/kg (N=9)
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Advate Dose Level: 25 IU/kg (N=7) | Advate Dose Level: 65 IU/kg (N=9) | BIVV001 Dose Level: 25 IU/kg (N=6) | BIVV001 Dose Level: 65 IU/kg (N=9)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Coagulation test abnormal (Investigations) | 1 | 0 | 0 | 0
Fibrin d dimer increased (Investigations) | 0 | 1 | 0 | 1
Thrombin-antithrombin iii complex increased (Investigations) | 1 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT03205163/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT03205163/SAP_001.pdf